CLINICAL TRIAL: NCT06501378
Title: Cranial Radiotherapy Plus PD-1/PD-L1 Inhibitors and Chemotherapy in Untreated Driver-mutation Negative Non-small Cell Lung Cancer With Active Brain Metastasis (BRILLIANT-1)
Brief Title: Cranial Radiotherapy Plus Chemoimmunotherapy in Untreated Driver-mutation Negative NSCLC With Active Brain Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024Lung-PD1-active BM
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- active BM (Experimental)
  Interventions: Drug: PD-1/PD-L1 inhibitor plus chemotherapy; Radiation: SRT/WBRT

INTERVENTIONS:
Drug: PD-1/PD-L1 inhibitor plus chemotherapy — Active brain metastases patients will receive PD-L1/PD-1 inhibitors and chemotherapy.
Radiation: SRT/WBRT — Active brain metastases (BM) patients will receive stereotactic radiotherapy (SRT) and whole brain radiation therapy (WBRT) according to their BM condition.

SUMMARY:
Non-small cell lung cancer (NSCLC), the most prevalent form of lung cancer, has a significant risk of brain metastasis (BM). Historically, the median overall survival for advanced NSCLC patients with BM was under six months with traditional chemotherapy. However, recent advancements with immune checkpoint inhibitors (ICIs) have shown promise, with some studies reporting improved intracranial objective response rates, progression-free survival, and overall survival when combined with chemotherapy.

Despite these improvements, challenges remain, such as treatment resistance, recurrence, and the need for better therapeutic strategies. Local interventions like stereotactic radiotherapy (SRT) and whole brain radiation therapy (WBRT) have been crucial for treating BM, with SRT being particularly effective. The combination of immunotherapy and radiotherapy is emerging as a synergistic approach, with studies suggesting it may enhance local control and survival rates while maintaining safety.

Guidelines recommend SRT for patients with limited BMs, and clinical data support the safety and efficacy of combining brain radiotherapy with immunotherapy. A meta-analysis and other studies have shown promising results with this combination, including local control rates and overall survival benefits, with manageable toxicities.

However, there is still a need for more prospective clinical trials to verify the safety and efficacy of combining cranial radiotherapy with immunotherapy in NSCLC patients with BM, especially those without driver gene mutations. Therefore, we plan to conduct a phase 2 prospective study, focusing on combining brain radiotherapy with PD-1/PD-L1 inhibitors. Though most of the current studies excluded patients with active BM, we believe that these patients need more attention. In this trial, we focus on patients with active BM and treat them with PD-1/PD-L1 inhibitor, chemotherapy and SRT/WBRT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* KPS score ≥ 70;
* Negative genetic testing for common driver genes including EGFR, ALK, ROS-1;
* Pathologically confirmed non-small cell lung cancer;
* Clinical stage IV (AJCC, 8th edition, 2017);
* Diagnosed with brain metastasis at the time of diagnosis, with at least one lesion in the brain with a diameter greater than 5mm on thin-section brain MRI;
* Active BMs that could not be controlled by symptomatic treatment, such as mannitol and dexamethasone
* Complete baseline assessment of systemic lesions before treatment, including enhanced brain MRI;
* Informed consent from the patient.

Exclusion Criteria:

* Multiple primary or metastatic tumors (except early skin cancer, cervical carcinoma in situ that has been treated radically, with no recurrence or progression for more than 5 years);
* Severe autoimmune diseases: active inflammatory bowel disease (including Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener's granulomatosis), etc.;
* Patients judged by the researcher as unsuitable for brain MRI or stereotactic brain radiotherapy;
* EGFR, ALK, or ROS1 gene mutations;
* Uncontrolled epilepsy, central nervous system disease, or history of mental disorders, judged by the researcher to potentially interfere with the signing of the informed consent form or affect patient compliance;
* Symptomatic interstitial lung disease or active infection/non-infectious pneumonia;
* Patients with risk factors for intestinal perforation: active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal cancer, or other known risk factors for intestinal perforation;
* Patients with active infection, heart failure, myocardial infarction within 6 months, unstable angina, or unstable arrhythmia;
* Other uncontrollable diseases or findings from physical examination or clinical experiments judged by the researcher to potentially interfere with the results or increase the risk of treatment complications for the patient;
* Mixed with small cell lung cancer components;
* Pregnant or lactating women;
* Congenital or acquired immunodeficiency diseases including HIV, or history of organ transplantation, allogeneic stem cell transplantation;
* Known HBV, HCV, active pulmonary tuberculosis infection;
* Patients who have received tumor vaccines, or have been vaccinated with other vaccines within 4 weeks before starting treatment (Note: Seasonal influenza vaccines are usually inactivated vaccines and are allowed, while nasal preparations are usually attenuated live vaccines and are not allowed);
* Concurrent use of other immunomodulators, chemotherapy drugs, drugs in other clinical studies, and long-term use of corticosteroid treatment are not eligible for inclusion;
* Patients allergic or contraindicated to PD-1/PD-L1 inhibitors or chemotherapy drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 1 year
  The time from the start of treatment until death from any cause. Patients who are still alive at the time of analysis will have their last contact date used as the cutoff date.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
  The percentage of participants who achieve a Complete Response (CR) or Partial Response (PR) after treatment, assessed according to the RECIST 1.1 criteria.
Intracranial Progression-Free Survival (iPFS) | 1 year
  The time from the start of treatment when the patient is enrolled until the observation of intracranial disease progression (appearance of new lesions, enlargement of existing lesions, excluding the possibility of pseudo-progression such as radiation necrosis) or death from any cause. Patients who have not progressed at the time of analysis will have their last contact date used as the cutoff date.
Intracranial Objective Response Rate (iORR) | 1 year
  The percentage of participants in the analysis population whose brain lesions achieve CR or PR, assessed according to the modified RECIST 1.1 criteria.
Progression-Free Survival (PFS) | 1 year
  The time from the start of treatment until the observation of disease progression or death from any cause, assessed according to the RECIST 1.1 criteria. Patients who are still alive at the time of analysis will have their last contact date used as the cutoff date.
Treatment-Related Adverse Event (TRAE) | 1 year
  Adverse events related to treatment, as assessed by the researcher, are recorded and evaluated according to the Common Terminology Criteria for Adverse Events(CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China